CLINICAL TRIAL: NCT04739696
Title: Cancer Caregivers and Their Struggle(s) Between Work and Family
Brief Title: Developing a Virtual Stress Management Intervention for Spousal/Partnered Caregivers of Solid Tumor Cancer Patients.
Acronym: eCare
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-2458.cc; 5R01CA231387-02 (NIH)
Record Dates: First submitted 2021-01-22; First posted 2021-02-05 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Lung Cancer; Colon Cancer; Solid Tumor, Adult
Keywords: depression; stress; caregiving; anxiety; psychoeducation intervention; psycho-oncology
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Colonic Neoplasms; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Caregiver Control (No Intervention): biomarker analysis; questionnaire administration; survey administration; treatment as usual
- Caregiver Intervention (Experimental): biomarker analysis; questionnaire administration; survey administration; PsychoEducation Paced Respiration and Relaxation (PEPRR), which includes virtual one-on-one psychoeducation and stress management intervention.
  Interventions: Behavioral: PEPRR
- Caregiver Self-Directed (Experimental): biomarker analysis; questionnaire administration; survey administration; Pep-Pal web-accessible video modules of the psychoeducation and stress management intervention.
  Interventions: Behavioral: Pep-Pal

INTERVENTIONS:
Behavioral: PEPRR — Briefly presented in the following order, sessions will include: 1) Overview and Introduction to Stress Management 2) Stress and the mind-body connection, 3) How our thoughts can lead to stress, 4) Coping with work and caregiver stress, 5) Strategies for maintaining energy and stamina with caregiver and work demands, 6) Coping with uncertainty and fear of unknown, 7) Managing changing relationships/communicating needs to employers and your loved ones, and 8) Getting the support they need including work accommodations and/or legal protections (e.g., Family Medical Leave Act, Americans with Disabilities Act)
  Other Names: Virtual-PEPRR; PsychoEducation Paced Respiration and Relaxation
  Arms: Caregiver Intervention
Behavioral: Pep-Pal — Pep-Pal program consisted of 11 sessions: 1) Introduction to stress management, 2) Stress and the mind body connection, 3) How thoughts can lead to stress, 4) Coping with stress, 5) Strategies for maintaining energy and stamina, 6) Coping with uncertainty, 7) Managing changing relationships and communicating needs, 8) Getting the support they need; 9) Employment related challenges and resources for working caregivers; 10) Employment session one; 11) Employment session two
  Arms: Caregiver Self-Directed

SUMMARY:
This randomized control trial will investigate the ability of an effective stress management psychoeducation program for employed caregivers to mitigate psychological distress and pathophysiology in spousal or partnered caregivers of patients' diagnosis with a solid tumor cancer of any stage. It is expected that improving caregiver status will have reduced depressive symptoms.

DETAILED DESCRIPTION:
Specific Aims

* Evaluate the impact of PsychoEducation Paced Respiration and Relaxation (PEPRR) delivered remotely as Virtual-PEPRR or online as Pep-Pal on caregivers employed at the time of their patient's cancer diagnosis and preselected based on high self-reported distress.
* Evaluate patient psychological status and healthcare utilization in patients whose caregivers received Virtual-PEPRR or Pep-Pal versus TAU
* Evaluate whether caregivers employment outcomes are associated with patient symptom management as an exploratory question.

OUTLINE: Caregivers are randomized to one of 3 groups (1:1:1) 1) Treatment as usual (TAU), 2) Virtual-PEPRR, or 3) Pep-Pal.

* Group I (treatment as usual [TAU]): Caregivers randomized to TAU will not participate in the stress management interventions. The TAU condition for this study takes into account published recommendations for an adequate representation of TAU. All participants regardless of randomization will be encouraged to use available psychological resources.
* Group II (Virtual PsychoEducation Paced Respiration and Relaxation [Virtual-PEPRR]): Caregivers participating in the Virtual-PEPRR intervention will consist of eight 60-75 minute video or telephone sessions. Each Virtual-PEPRR session will be devoted to a specific topic with the goal of assisting the caregiver in developing and applying stress-management skills both in caregiving as well as in their work setting. Sessions include problem-solving, identifying cognitive distortions, application of relaxation techniques such as the emWave2, acquiring new coping skills, utilizing social support, and establishing appropriate goals, and finding support. All caregivers in Virtual-PEPRR will be provided a Caregiver Workbook that includes information about the session topics and homework assignments.
* Group III (Pep-Pal): Pep-Pal is a mobilized version of Virtual-PEPRR. Pep-Pal includes eleven web-based video modules replicate essential components of each session of Virtual-PEPRR, but in shorter format (<20 minute. duration) with engaging relaxation exercises. The modules include learning skills in problem-solving, identifying cognitive distortions, using relaxation techniques, acquiring new coping skills, utilizing social support, establishing suitable goals, and finding support. Pep-Pal includes "Mini-Peps" which are video guided, 3-minute stress reduction exercises that the caregiver can access any time. Caregivers randomized to Pep-Pal will complete modules at times that are convenient and web-accessible by smartphone, tablet, laptop, or desktop computer. Caregivers can complete more than one module a week, repeat any session, and access the Mini-Peps as frequently as desired.

Caregivers and patients undergo psychosocial assessments prior to randomization, and at 3 months, 6 months, 9 months and 1 year after baseline. At each phase, caregivers and patients will complete battery of questionnaires that includes the Center for Epidemiological Studies-Depression scale (CES-D), the perceived stress scale (PSS), and the State-Trait Anxiety Inventory (STAI). Caregivers will be asked monthly to complete eight very short questions Patient-Reported Outcomes Measurement Information System (PROMIS). Additionally the patient will complete the MD Anderson Symptom Inventory each time while the caregiver completes questionnaires will cover details about how being a caregiver has affected their lives, details about employment, insurance and accommodations, general physical and mental well-being, and the impact Covid-19 has had on their lives. The patient and the caregiver will additionally complete a demographic questionnaire that includes questions regarding age, diagnosis, income, and other standard questions regarding nutrition, health behaviors, and health services utilization. At study completion, an exit questionnaire will address each subject's evaluation of the study and the group in which they were assigned.

Saliva and hair samples from caregivers will be collected every three months: baseline, 3 months, 6 months, 9 months and 1 year after baseline.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS (Meets all of the following criteria):

Patients who have a primary diagnosis of solid tumor cancer at any stage that are within 12 weeks +/- of starting treatment, which includes either infusion chemo- or immunotherapy, oral targeted agents, or both.

PATIENT CHARACTERISTICS:

* Patients who have a primary diagnosis of soled tumor cancer at any stage that are within 12 weeks of initiating treatment.
* Patient must be spouse or partner of the caregiver for at least a year and must live with caregiver
* Must be able to read/speak English
* 18 years of age or older

CAREGIVER CHARACTERISTICS:

* A primary caregiver for the patient with a diagnosis of solid tumor cancer at any stage who are within 12 weeks of initiating treatment
* Spouse or partner of the patient for at least a year
* The caregiver must live with the patient
* Must be available to fully participate in an intervention (Virtual-PEPRR or PepPal) if assigned
* Must score 1 or greater on the PHQ-2 (depression) and/or GAD-2 (anxiety) during pre-screening.
* Must be employed at the time of the patient's diagnosis for a minimum of 20 hours/week with plans to remain employed and working during their patient's treatment. Caregivers that were furloughed or laid off due to Covid-19 who are actively looking for work will be included.
* Able to read and speak the English language
* Willingness to use a Smartphone
* Age 25 (inclusive) 65 (non-inclusive)

Exclusion Criteria:

* Having a serious medical condition likely to influence neuroendocrine parameters
* Chronic use of steroid medications
* If Female, pregnant or planning to become pregnant in the next year
* History of a psychiatric illness unrelated to their experience as a caregiver with the past 18 months.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 510 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Caregiver: Change in Center for Epidemiological Studies Depression Scale (CESD) | Baseline, 3 months, 6 months, 9 months, 12 months follow up
  Change in caregiver depressive symptoms. Center for Epidemiological Studies Depression Scale (CESD) is a self-report 20-item scale designed to measure current depressive symptoms. Total score range from 0-60, with a score at or above 16 reflecting significant depressive symptomatology.

SECONDARY OUTCOMES:
Caregiver: Change in Spielberger State-Trait Anxiety Inventory (STAI) | Baseline, 3 month, 6 month, 9 month, 12 month follow up
  Change in caregiver anxiety. The "Spielberger State and Trait Anxiety Inventory" (STAI) is a validated self-reporting instrument used to assess anxiety in adults. The inventory consists of state anxiety, which evaluates how the subject feels currently (transient anxiety). The scale consists of 20 questions, and a higher score indicates greater anxiety. Total score ranges from 20 (no anxiety) to 80 (maximum anxiety).
Caregiver: Change in Perceived Stress Scale (PSS) | Baseline, 3 month, 6 month, 9 month, 12 month follow up
  Change in caregiver perceived stress. The "Perceived Stress Scale" (PSS) measures the overall level of stress. This instrument contains 14 items accessing overall appraisals of stress in the past month. The total score range is 0-56. A higher score indicates greater stress.
Caregiver: Health Care Utilization | Baseline, 12 month follow up
  Caregiver electronic health records and supplemented by Colorado All Payer Claims Data and self-report
Caregiver: Change in Adrenal Activity Over Time | Baseline, 3 month, 6 month, 9 month, 12 month follow up
  Cortisol measured in hair will be used as a retrospective measure of activation of the hypothalamic pituitary adrenal axis.
Caregiver: Change in Caregiver Telomere Length Over Time | Baseline, 3 month, 6 month, 9 month, 12 month follow up
  Telomere length was assessed as a measure of cellular aging in blood samples from participants.
Patient: Change in Center for Epidemiological Studies Depression Scale (CESD) | Baseline, 3 month, 6 month, 9 month, 12 month follow up
  Change in patient depressive symptoms. Center for Epidemiological Studies Depression Scale (CESD) is a self-report 20-item scale designed to measure current depressive symptoms. Total score range from 0-60, with a score at or above 16 reflecting significant depressive symptomatology.
Patient: Change in Spielberger State-Trait Anxiety Inventory (STAI) | Baseline, 3 month, 6 month, 9 month, 12 month follow up
  Change in patient anxiety. The "Spielberger State and Trait Anxiety Inventory" (STAI) is a validated self-reporting instrument used to assess anxiety in adults. The inventory consists of state anxiety, which evaluates how the subject feels currently (transient anxiety). The scale consists of 20 questions, and a higher score indicates greater anxiety. Total score ranges from 20 (no anxiety) to 80 (maximum anxiety).
Patient: Change in Perceived Stress Scale | Baseline, 3 month, 6 month, 9 month, 12 month follow up
  Change in patient perceived stress. The "Perceived Stress Scale" (PSS) measures the overall level of stress. This instrument contains 14 items accessing overall appraisals of stress in the past month. The total score range is 0-56. A higher score indicates greater stress.
Patient: Health Care Utilization | Baseline, 12 month follow up
  Patient electronic health records and supplemented by Colorado All Payer Claims Data
Patient: Change in MD Anderson Symptom Inventory (MDASI) | Baseline, 3 month, 6 month, 9 month, 12 month follow up
  Patient symptom management. the MD Anderson Symptom Inventory (MDASI) core scale, which assesses 13 symptoms (pain, fatigue, nausea, disturbed sleep, distress, shortness of breath, memory problems, lack of appetite, drowsiness, dry mouth, numbness, sadness, and vomiting) on a 0-10 scale.
Caregiver: Employment status | Baseline, 12 month follow up
  Caregiver self-report employment and weekly hours worked questions from Current Population Survey (CPS)
Caregiver: Job Satisfaction | Baseline, 12 month follow up
  Caregiver self-report job satisfaction. Job satisfaction is measured by a single-item assessment tool assessing whether or not the participant was satisfied with their current job. Satisfaction was measured on a 0-7 scale. Higher score indicates a higher level of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Cathy J Bradley, PhD, Principal Investigator — University of Colorado Denver (Anschutz Medical Campus)
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States